CLINICAL TRIAL: NCT06073938
Title: A Real-World Study of NHWD-870 in Patients With Advanced Solid Tumors or Lymphomas Carrying NUT Rearrangement
Brief Title: Compassionate Use Study of NHWD-870 in Patients With Advanced Solid Tumors or Lymphomas Carrying NUT Rearrangement
Status: Recruiting | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Deputy Director of Thoracic Oncology Department, Hunan Province Tumor Hospital
Other Study IDs: BRD-870 RWS
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumors or Lymphomas
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples，tumor tissue samples (by puncture, incision or clamping)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: NHWD-870 — The base dosage administered is 2.0 mg/dose/day, and the frequency and dose of administration may be adjusted based on safety data.

SUMMARY:
The NHWD-870 Phase I clinical trial evaluated the safety, tolerability, pharmacokinetics and pharmacodynamics in patients with advanced tumors. The objectives of this retrospective study were to preliminarily evaluate the anti-tumor efficacy of NHWD-870 HCl in patients with advanced solid tumors or lymphomas and to preliminarily evaluate biomarkers associated with the efficacy of NHWD-870 HCl in the treatment of patients with advanced solid tumors or lymphomas, to provide a basis for identifying the enriched population for the late-stage trial.

ELIGIBILITY:
Inclusion Criteria:

1. Signing an informed consent form;
2. Patients with advanced solid tumors or lymphomas definitively diagnosed by pathology;
3. Age ≥18 and ≤75 years;
4. Eastern Cooperative Oncology Group (ECOG) score physical status score of 0 to 1;
5. Expected survival of >3 months;
6. NUT positive confirmed by molecular testing.

Exclusion Criteria:

Subjects who meet one or more of the following criteria will be excluded:

1. Other serious complications (such as uncontrolled infection, myocardial infarction within 6 months, high blood pressure (≥ 160/100mmHg) and thromboembolic disease that cannot be controlled by drug intervention, etc.);
2. The adverse reactions of previous anti-tumor therapy have not been restored to CTCAE 5.0 ≤ Grade1 (except for hair loss, anemia and other toxicities judged by researchers to be unsafe);
3. History of substance abuse;
4. Inability to take drugs due to dysphagia (except for patients who receive nutrients through a gastric tube due to dysphagia), or conditions that the investigator determines seriously affect gastrointestinal absorption;
5. Patients with a history of other serious systemic diseases who are judged by the investigator to be unsuitable for participating in clinical trials;
6. Alcoholics or those who drink more than 28 units of alcohol per week (1 unit = 285 mL of beer or 25 mL of spirits or 1 glass of wine);
7. Suffering from uncontrollable mental illness;
8. Pregnant or lactating women, or patients of childbearing age (including male subjects) with pregnancy plans;
9. Active hepatitis B (viral titer >103), hepatitis C or HIV ( );
10. Long-term treatment with high-dose corticosteroids or other immunosuppressants, such as those who have undergone organ transplantation, or those who have received systemic glucocorticoids (such as prednisone> 10 mg/day or equivalent drugs) or other immunosuppressant therapy within 14 days before the first use of the study drug; Exceptions are given for topical, ocular, intra-articular, intranasal and inhaled corticosteroid therapy; short-term use of glucocorticoids for prophylaxis (e.g., prevention of contrast allergy);
11. The investigator believes that the subject is not suitable to participate in this clinical study for other objective reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced solid tumors or lymphomas, NUT rearrangement positive
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 1.5 years
  Proportion of patients whose tumor volume shrinks to a pre-specified value (usually 30%) and who are able to maintain the minimum timeframe requirements.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincal Tumor Hospital, Changsha, Hunan, China